CLINICAL TRIAL: NCT06707727
Title: Characteristics and Prognostic Outcomes of Diaphragmatic Ultrasound in Myasthenia Gravis
Status: Active, not recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Fei Xiao, Prof.Fei Xiao, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2024-050-01
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Myasthaenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- myasthenia gravis
- controls

SUMMARY:
The goal of this observational study is to learn about the characteristics and prognostic outcomes of diaphragmatic ultrasound in myasthenia gravis. The main question it aims to answer is:

Does diaphragmatic ultrasound predict prognosis of myasthenia gravis in six months? Participants diagnosed as myasthenia gravis will take the diaphragm ultrasound examinations.

ELIGIBILITY:
Inclusion Criteria:

* 1: Patients who seek treatment at the First Affiliated Hospital of Chongqing Medical University and have fluctuating skeletal muscle weakness and at least one of the following three conditions will be included: positive reaction to cholinesterase inhibitors

  2: Serum positive antibodies against acetylcholine receptors, muscle specific kinases, or lipoprotein related proteins

  3: Repeated electrical stimulation examination showed a decrease in wave amplitude.

Exclusion Criteria:

* 1: Patients with lung disease or heart failure, or a history of non-invasive ventilator or tracheotomy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who seek treatment at the First Affiliated Hospital of Chongqing Medical University and have fluctuating skeletal muscle weakness and at least one of the following three conditions will be included: positive reaction to cholinesterase inhibitors; Serum positive antibodies against acetylcholine receptors, muscle specific kinases, or lipoprotein related proteins; Repeated electrical stimulation examination showed a decrease in wave amplitude.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
QMG changes | 6 months

SECONDARY OUTCOMES:
Changes in medication type or dose | 6 months
  acetylcholinesterase inhibitors, glucocorticoid, immunosuppressant
respiratory infection | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes